CLINICAL TRIAL: NCT05454995
Title: Feasibility Study of the Vessel Restoration System (VRS) for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA): ACTIVATE II
Brief Title: Feasibility Study of the Vessel Restoration System (VRS): ACTIVATE II
Acronym: ACTIVATEII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alucent Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1061-001
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: PAD - Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: NVS Therapy will be delivered to de novo lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) during PTA in patients with symptomatic peripheral artery disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Alucent VRS for Treatment of Atherosclerotic Lesions (Experimental): Combination Product: VRS
  Interventions: Other: Vessel Restoration System (VRS)

INTERVENTIONS:
Other: Vessel Restoration System (VRS) — Vessel Restoration System (VRS) for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA)

SUMMARY:
Feasibility Study of the Vessel Restoration System (VRS) for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA): ACTIVATE II

ELIGIBILITY:
General Inclusion Criteria

1. Subject (or Legal Guardian) is willing and able to provide consent before any study-specific tests or procedures are performed and agree to attend all required follow-up visits.
2. Male or female subject of at least 18 years of age.
3. Chronic symptomatic lower limb ischemia defined as Rutherford classification 2, 3, or 4.

General Exclusion Criteria

1. Life expectancy, documented in the Investigator's opinion, of less than 1 year.
2. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) or cardiac event (e.g., PCI for STEMI/NSTEMI, unstable angina) within 6 months prior to the index procedure.
3. Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant/antiplatelet therapies.
4. Use of rivaroxaban 2.5 mg BID with low-dose aspirin for the treatment of patients with symptomatic peripheral arterial disease is permitted as per local standard of care. Use of rivaroxaban 2.5 mg in conjunction with dual antiplatelet therapy (low-dose aspirin and a secondary agent) is not permitted.
5. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated.
6. Chronic renal insufficiency with serum creatinine ≥2.5 mg/dL or eGFR <45 ml/min within 30 days prior to the index procedure or treatment with peritoneal or hemodialysis.
7. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3 within 30 days prior to the index procedure or has a history of bleeding diathesis.
8. Receiving oral or intravenous immunosuppressive therapy.
9. Subject is currently receiving a medication that causes photosensitivity, with a prior documented photosensitive reaction.
10. Subject has white blood cell (WBC) count <3.0 (3,000 cells/mm3) within 30 days prior to the index procedure.
11. Subject has known or suspected active systemic infection evidenced by WBC > 14.0 (14,000/mm3).
12. History of major amputation in the target limb.
13. Any major intervention planned at the index procedure or within 30 days post-index procedure including treatment of contralateral limb.
14. Any arterial access other than contralateral common femoral artery (CFA) or ipsilateral antegrade CFA is required to gain access to target vessel. All popliteal and infrapopliteal ipsilateral retrograde access are excluded.
15. Subject has any permanent neurologic defect that may impair ambulation and/or cause non-compliance with the protocol.
16. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding within 6 months prior to the index procedure.
17. Subject has documented or suspected liver disease, including laboratory evidence of hepatitis.
18. Subject is currently on oral anticoagulation therapy, such as warfarin, rivaroxaban, apixaban, or dabigatran etexilate, except when the subject is prescribed such medication as treatment for atrial fibrillation (medication and/or following ablation therapies and/or left atrial appendage occlusion procedure). Use of low-dose rivaroxaban 2.5 mg BID and low-dose aspirin to treat patients with symptomatic peripheral arterial disease is permitted as per local standard of care.
19. Subject is planned to undergo treatment with the ShockWave® IVL (ShockWave Medical Inc. Santa Clara, CA, USA) and/or any adjunctive pre-dilatation vessel preparation angioplasty device.
20. Subject is pregnant, breastfeeding, or planning to become pregnant in the next 30 days. Subjects (male and female) of childbearing potential must agree to use effective birth control measures for 30 days after the index procedure.
21. Current or planned (within one-year post-index procedure) participation in another investigational drug or device clinical trial that has not completed the primary endpoint at the time of randomization/enrollment or that clinically interferes with the current trial endpoints.
22. Any concurrent condition which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol and follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
To assess the safety | 12 months
  To assess the safety of the VRS by way of occurence of advese events during the index procedure
To assess efficacy | 12 months
  To assess the efficacy of the VRS as determined by lesion patency through 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Flinders Medical Center, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No